CLINICAL TRIAL: NCT04175808
Title: Single-dose and Randomized, Single-center, Placebo- and Active-controlled, Crossover Study to Assess the Effect of Omecamtiv Mecarbil (OM) on QT/QTc Intervals in Healthy Subjects
Brief Title: Study to Assess the Effect of Omecamtiv Mecarbil (OM) on QT/QTc Intervals in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cytokinetics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 20090231; 2018-003157-19 (EudraCT Number)
Record Dates: First submitted 2019-11-07; First posted 2019-11-25 (Actual); Results first posted 2021-07-20 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: QT Intervals Changes; QTc Intervals Changes
Keywords: Thorough QT; QTc study
MeSH Terms: interventions — omecamtiv mecarbil; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This was a partially double-blind study. In Part B, placebo and OM treatments were double-blinded, moxifloxacin treatment was open-label, and the core ECG laboratory was blinded to all treatment information. Except for the moxifloxacin treatment in 1 of 3 periods in Part B, treatment assignment was blinded to all participants, site personnel, the Medical Monitor, and Clinical Research Associates.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part A (Experimental): After an overnight fast of at least 10 hours participants received a single oral dose of 25 mg omecamtiv mecarbil on Day 1.
  Interventions: Drug: Omecamtiv Mecarbil (OM)
- Part B (Experimental): Participants with a maximum observed plasma OM concentration ≤ 350 ng/mL in Part A were randomly assigned to receive a single dose of each the following 3 treatments in one of six treatment sequences:
  * Placebo
  * 50 mg omecamtiv mecarbil
  * 400 mg moxifloxacin Each treatment was separated by a washout of at least 7 days.
  Interventions: Drug: Omecamtiv Mecarbil (OM); Drug: Placebo; Drug: Moxifloxacin

INTERVENTIONS:
Drug: Omecamtiv Mecarbil (OM) — Oral solution
  Other Names: AMG 423
Drug: Placebo — Placebo oral solution
  Arms: Part B
Drug: Moxifloxacin — 400 mg moxifloxacin oral tablet
  Arms: Part B

SUMMARY:
The primary objective of this study is to assess the effect of a single therapeutic (50 mg) oral dose of omecamtiv mecarbil (OM) on the QT interval / QT interval corrected for heart rate (QTc), relative to placebo, in healthy adults.

The QT interval is the section on an electrocardiogram (ECG) that represents the time it takes for the electrical system to fire an impulse through the ventricles and then recharge, or the time it takes for the heart muscle to contract and then recover.

DETAILED DESCRIPTION:
The study consists of 2 parts: Part A and Part B. Participants are enrolled in Part A to determine eligibility for Part B.

In Part A participants receive a single oral dose of 25 mg omecamtiv mecarbil; participants with a resulting maximum observed OM plasma concentration (Cmax) ≤ 350 ng/mL are eligible to enter Part B.

Part B is a 3-period cross-over study in which participants are randomized to receive 3 treatments in 1 of 6 sequences, each separated by a washout of at least 7 days.

This study was conducted by Amgen as the IND holder, with Cytokinetics as a collaborator. Due to the termination of the collaboration agreement between Amgen and Cytokinetics in May 2021 and subsequent transfer of the omecamtiv mecarbil IND from Amgen to Cytokinetics, Cytokinetics is now listed as the sponsor.

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided informed consent before initiation of any study-specific activities/procedures.
* Healthy male or healthy female subjects greater than or equal to 18 to less than or equal to 50 years of age.
* No history or evidence of clinically relevant medical disorders as determined by the Investigator at Screening.
* Physical examination at Screening and vital signs, clinical laboratory values, and electrocardiogram (ECG) at Screening and Day -1 of each period are clinically acceptable to the Investigator.
* Body mass index (BMI) greater than, or equal to 18.0 kg/m^2 and less than, or equal to 30.0 kg/m^2.
* Willing to maintain current general diet and physical activity regimen.

Exclusion Criteria:

* History or evidence of clinically significant disorder, condition, or disease not otherwise excluded that, in the opinion of the Investigator, would pose a risk to subject safety or interfere with the study evaluation, procedures, or completion.
* Any users of tobacco- or nicotine-containing products within 6 months before Day -1 of Part A.
* History suggestive of esophageal (including esophageal spasm, esophagitis), gastric, or duodenal ulceration or bowel disease (including, but not limited to, peptic ulceration, gastrointestinal bleeding, ulcerative colitis, Crohn's disease, or irritable bowel syndrome); or a history of gastrointestinal surgery other than uncomplicated appendectomy.
* History or current signs or symptoms of cardiovascular disease, including but not limited to myocardial infarction, congenital heart disease, valvular heart disease, coronary revascularization, or angina.
* Known substance abuse (eg, alcohol, licit or illicit drugs) within 1 year prior to Screening.
* Subjects with poor peripheral venous access.
* Use of any medications/substances outside the allowed timeframes as specified in Section 6.1.2.
* Currently receiving treatment in another investigational device or drug study, or less than 3 months, or 5 half-lives if longer, prior to receiving the first dose of study drug. Other investigational procedures while participating in this study are excluded.
* Donated blood from 3 months prior to Screening, plasma from 2 weeks prior to Screening, or platelets from 6 weeks prior to Screening.
* Subjects who were previously exposed to OM.
* Hepatic impairment defined by a total bilirubin (TBL) greater than or equal to 1.2 times the upper limit of normal (ULN), or alanine aminotransferase (ALT) or aspartate aminotransferase (AST) greater than ULN (and confirmed upon repeat).
* Systolic blood pressure (BP) greater than 140 mmHg or less than 90 mmHg, or diastolic BP greater than 90 mmHg.
* QTcF interval greater than 450 msec in male or greater than 470 msec in female or history/evidence of long QT syndrome, or PR of greater than or equal to 200 msec; or 2nd degree atrioventricular (AV) block or 3rd degree AV block, or heart rate greater than 100 bpm (and confirmed upon repeat, except 2nd or 3rd degree AV block, which are exclusionary based on a single finding).
* Troponin I or creatine kinase MB fraction (CK-MB) greater than ULN at Screening or Check-in for Part A or B.
* Estimated glomerular filtration rate (eGFR) less than 80 mL/min/1.73 m^2 at Screening as calculated by the Modified Diet in Renal Disease (MDRD) equation;
* Any positive test for drugs, cotinine (tobacco or nicotine use), and/or alcohol use.
* Positive hepatitis panel and/or positive human immunodeficiency virus test. Subjects whose results are compatible with prior immunization may be included.
* Subject has known sensitivity to any of the products or components to be administered during dosing, including history of hypersensitivity to moxifloxacin or any member of the quinolone class of antibacterials.
* History of tendon rupture or connective tissue disorders.
* Female subjects with a positive pregnancy test.
* Female subjects lactating/breastfeeding or who plans to breastfeed during the study through 90 days after the end of study (EOS) visit.
* Unwilling to adhere to contraceptive requirements through 90 days after the EOS visit.
* Unwilling to abstain from sperm and ovum donation through 90 days after the EOS visit.
* Male subjects with a female partner of childbearing potential and not willing to inform his partner of his participation in this clinical study.
* Male subjects with a pregnant partner or partner planning to become pregnant while the subject is on study through 90 days after the EOS visit.
* Subject likely to not be available to complete all protocol-required study visits or procedures, and/or to comply with all required study procedures (eg, Clinical Outcome Assessments) to the best of the subject and Investigator's knowledge.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2019-11-14 (Actual); Primary Completion 2020-03-04 (Actual); Study Completion 2020-03-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (1):
- Research Site, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at a single site in the United Kingdom. The study consisted of 2 parts: Part A and Part B.
  Part A was a lead-in phase to ensure that omecamtiv mecarbil (OM) plasma concentrations in Part B would not exceed 1000 ng/mL.
Pre-assignment Details: Participants in Part A received a single oral dose of 25 mg omecamtiv mecarbil; participants with maximum observed OM plasma concentration (Cmax) ≤ 350 ng/mL were eligible to enter Part B.
  Part B was a 3-period cross-over study in which all participants received a single dose of placebo, omecamtiv mecarbil, and moxifloxacin in 1 of 6 sequences, each separated by a washout of at least 7 days.
Groups:
- Part B: Placebo/OM/Moxifloxacin: Participants received a single dose of placebo oral solution in Period 1, 50 mg omecamtiv mecarbil oral solution in Period 2 and 400 mg moxifloxacin oral tablet in Period 3. Each treatment was separated by a washout period of at least 7 days.
- Part B: OM/Moxifloxacin/Placebo: Participants received a single dose of 50 mg omecamtiv mecarbil oral solution in Period 1, 400 mg moxifloxacin oral tablet in Period 2, and placebo oral solution in Period 3. Each treatment was separated by a washout period of at least 7 days.
- Part B: Moxifloxacin/Placebo/OM: Participants received a single dose of 400 mg moxifloxacin oral tablet in Period 1, placebo oral solution in Period 2, and 50 mg omecamtiv mecarbil oral solution in Period 3. Each treatment was separated by a washout period of at least 7 days.
- Part B: Placebo/Moxifloxacin/OM: Participants received a single dose of placebo oral solution in Period 1, 400 mg moxifloxacin oral tablet in Period 2, and 50 mg omecamtiv mecarbil oral solution in Period 3. Each treatment was separated by a washout period of at least 7 days.
- Part B: Moxifloxacin/OM/Placebo: Participants received a single dose of 400 mg moxifloxacin oral tablet in Period 1, 50 mg omecamtiv mecarbil oral solution in Period 2, and placebo oral solution in Period 3. Each treatment was separated by a washout period of at least 7 days.
- Part B: OM/Placebo/Moxifloxacin: Participants received a single dose of 50 mg omecamtiv mecarbil oral solution in Period 1, placebo oral solution in Period 2, and 400 mg moxifloxacin oral tablet in Period 3. Each treatment was separated by a washout period of at least 7 days.
Period: Part A
Arm/Group | Part A | Part B: Placebo/OM/Moxifloxacin | Part B: OM/Moxifloxacin/Placebo | Part B: Moxifloxacin/Placebo/OM | Part B: Placebo/Moxifloxacin/OM | Part B: Moxifloxacin/OM/Placebo | Part B: OM/Placebo/Moxifloxacin
Started | 70 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 68 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Miscellaneous | 2 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part B
Arm/Group | Part A | Part B: Placebo/OM/Moxifloxacin | Part B: OM/Moxifloxacin/Placebo | Part B: Moxifloxacin/Placebo/OM | Part B: Placebo/Moxifloxacin/OM | Part B: Moxifloxacin/OM/Placebo | Part B: OM/Placebo/Moxifloxacin
Started | 0 | 10 | 10 | 10 | 10 | 10 | 10
Completed | 0 | 10 | 10 | 10 | 10 | 10 | 10
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants randomized in Part B of the study
Groups:
- Part B: Participants with a maximum observed OM plasma concentration ≤ 350 ng/mL in Part A were randomly assigned to receive a single dose of each the following 3 treatments in one of six treatment sequences:
  * Placebo
  * 50 mg omecamtiv mecarbil
  * 400 mg moxifloxacin Each treatment was separated by a washout of at least 7 days.
Arm/Group | Part B
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.7 (8.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 60
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 49
  Black or African American | 6
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  American Indian or Alaska Native | 0
  Multiple | 1
QT Interval Corrected for Heart Rate Based on the Fridericia Method (QTcF) [Mean (Standard Deviation); unit: ms] — In Part B, continuous 12-lead digital electrocardiogram (ECG) recording was performed on Day 1 of each treatment period. Up to 10 digital 12-lead ECG tracings were extracted at -1.25, -1, and -0.75 hours pre-dose. The median QTc value from all beats in each replicate was calculated and then the mean of the available medians was used as the participant's reportable value at that time point. Baseline was the average of the values from the 3 pre-dose time points (-1.25, -1, and -0.75 hours) on Day 1 for the respective treatment period.
  ms
    Prior to OM dose | 402.9 (18.27)
    Prior to moxifloxacin dose | 402.4 (18.38)
    Prior to placebo dose | 404.1 (19.06)
PR Interval [Mean (Standard Deviation); unit: ms] — The PR interval is the time from the onset of the P-wave to the start of the next QRS complex.
  ms
    Prior to OM dose | 151.4 (22.48)
    Prior to moxifloxacin dose | 150.7 (22.73)
    Prior to placebo dose | 151.2 (24.20)
QRS [Mean (Standard Deviation); unit: ms] — The QRS complex is a combination of the Q wave, R wave and S wave on an ECG tracing, and represents ventricular depolarization.
  ms
    Prior to OM dose | 105.6 (5.74)
    Prior to moxifloxacin dose | 105.8 (5.36)
    Prior to placebo dose | 105.8 (5.52)
Heart Rate [Mean (Standard Deviation); unit: beats/minute]
  Prior to OM dose | 59.2 (7.87)
  Prior to moxifloxacin dose | 59.5 (7.36)
  Prior to placebo dose | 58.6 (8.03)

OUTCOME MEASURES:

1. Primary Outcome: Placebo-corrected Change From Baseline in QT Interval Corrected for Heart Rate Based on the Fridericia Method (QTcF) After Omecamtiv Mecarbil Dosing in Part B
Description: Continuous 12-lead digital ECG recording was performed on day 1 of each period. ECGs were analyzed by a blinded, central reader. At each specified timepoint, ten 14-second 12-lead ECG tracings were extracted from the continuous recordings. The median QT in each replicate was calculated; the mean of available medians was used as the participant's reportable value at that timepoint.
  QT interval was corrected for heart rate using Fridericia's correction (QTcF). Change from baseline (ΔQTcF) was calculated based on a linear mixed-effects model with period, sequence, time (categorical), treatment, and time-by-treatment interaction as fixed effects and baseline QTcF as covariate.
  Placebo-corrected ΔQTcF (ΔΔQTcF) was calculated as the adjusted mean ΔQTcF after OM dosing minus adjusted mean ΔQTcF after placebo.
  If the upper bound of the confidence interval of ΔΔQTcF was < 10 ms for all post-dose time points, OM was to be concluded to not have a significant effect on QT interval prolongation.
Time Frame: Baseline (average of samples taken at -1.25, -1, and -0.75 hours predose on day 1 of the treatment period) and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 8, 12, and 24 hours post-dose
Population: The QT/QTc analysis set included all participants who received at least 1 dose of study treatment with measurements at baseline as well as on-treatment with at least 1 postdose timepoint with a valid ΔQTcF value in Part B.
Measure: Least Squares Mean (90% Confidence Interval); unit: ms
Groups:
- Part B: Omecamtiv Mecarbil 50 mg: Participants received a single oral dose of 50 mg OM on day 1 of treatment period 1, 2, or 3, depending on sequence assignment.
Arm/Group | Part B: Omecamtiv Mecarbil 50 mg
Number analyzed (Participants) | 60
ms
  0.25 hours post-dose | -2.6 [-3.87 to -1.24]
  0.5 hours post-dose | -4.9 [-6.40 to -3.45]
  0.75 hours post-dose | -5.8 [-7.34 to -4.18]
  1 hour post-dose | -6.7 [-8.13 to -5.29]
  1.5 hours post-dose | -4.5 [-5.95 to -2.98]
  2 hours post-dose | -2.7 [-4.21 to -1.18]
  3 hours post-dose | -1.5 [-2.96 to -0.10]
  4 hours post-dose | -0.8 [-2.35 to 0.70]
  8 hours post-dose | -2.2 [-4.10 to -0.24]
  12 hours post-dose | -1.9 [-3.98 to 0.22]
  24 hours post-dose | -1.2 [-2.68 to 0.30]

2. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Omecamtiv Mecarbil in Part B
Description: Plasma samples at each timepoint were quantified using a validated liquid chromatography-tandem mass spectrometry method. The lower limit of quantification for plasma samples was 1 ng/mL.
Time Frame: Day 1 of the OM treatment period at pre-dose and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 8, 12, 24, 48, 72, 96, and 120 hours post-dose.
Population: The pharmacokinetic (PK) population for Part B consisted of all participants who received OM and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part B: Omecamtiv Mecarbil 50 mg
Number analyzed (Participants) | 60
ng/mL | 416 (33.2)

3. Secondary Outcome: Time to Maximum Observed Plasma Concentration (Tmax) of Omecamtiv Mecarbil In Part B
Time Frame: as for outcome 2
Population: Part B PK population
Measure: Median (Full Range); unit: hours
Arm/Group | Part B: Omecamtiv Mecarbil 50 mg
Number analyzed (Participants) | 60
hours | 0.583 [0.333 to 1.08]

4. Secondary Outcome: Apparent Terminal Elimination Half-life (T1/2) of Omecamtiv Mecarbil in Part B
Time Frame: as for outcome 2
Population: Part B PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Part B: Omecamtiv Mecarbil 50 mg
Number analyzed (Participants) | 60
hours | 20.0 (2.91)

5. Secondary Outcome: Apparent Total Plasma Clearance (CL/F) for Omecamtiv Mecarbil in Part B
Time Frame: as for outcome 2
Population: Part B PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Part B: Omecamtiv Mecarbil 50 mg
Number analyzed (Participants) | 60
L/h | 10.4 (21.2)

6. Secondary Outcome: Apparent Volume of Distribution (VZ/F) for Omecamtiv Mecarbil in Part B
Time Frame: as for outcome 2
Population: Part B PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | Part B: Omecamtiv Mecarbil 50 mg
Number analyzed (Participants) | 60
liters | 299 (21.5)

7. Secondary Outcome: Area Under the Concentration-time Curve From Time 0 to the Time of Last Quantifiable Concentration (AUC0-t) for Omecamtiv Mecarbil in Part B
Time Frame: as for outcome 2
Population: Part B PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part B: Omecamtiv Mecarbil 50 mg
Number analyzed (Participants) | 60
h*ng/mL | 4710 (21.0)

8. Secondary Outcome: AUC From Time 0 to Infinity (AUCinf) for Omecamtiv Mecarbil in Part B
Time Frame: as for outcome 2
Population: Part B PK population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part B: Omecamtiv Mecarbil 50 mg
Number analyzed (Participants) | 60
h*ng/mL | 4790 (21.2)

9. Secondary Outcome: Placebo-corrected Change From Baseline in QT Interval Corrected for Heart Rate Based on the Fridericia Method (QTcF) After Moxifloxacin Dosing in Part B
Description: Assay sensitivity was validated by analysis of ∆QTcF of moxifloxacin. Continuous 12-lead digital ECG recording was performed on Day 1 of each period. ECGs were analyzed by a blinded, central reader. At each specified timepoint, ten 14-second 12-lead ECG tracings were extracted from the continuous recordings. The median QT in each replicate was calculated; the mean of available medians was used as the participant's reportable value at that timepoint.
  QT interval was corrected for heart rate using Fridericia's correction (QTcF). Change from baseline (ΔQTcF) was calculated based on a linear mixed-effects model with period, sequence, time (categorical), treatment, and time-by-treatment interaction as fixed effects and baseline QTcF as covariate.
  Placebo-corrected ΔQTcF (ΔΔQTcF) was calculated as the adjusted mean ΔQTcF after moxifloxacin dosing minus adjusted mean ΔQTcF after placebo.
  If ∆∆QTcF was larger than 5 ms at 2, 3, or 4 hours, assay sensitivity was considered to be demonstrated.
Time Frame: Baseline (average of samples taken at -1.25, -1, and -0.75 hours predose on day 1 of the moxifloxacin treatment period) and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 8, 12, and 24 hours post-dose.
Population: The QT/QTc analysis set
Measure: Least Squares Mean (90% Confidence Interval); unit: ms
Groups:
- Part B: Moxifloxacin 400 mg: Participants received a single dose of 400 mg moxifloxacin on day 1 of treatment period 1, 2, or 3, depending on sequence assignment.
Arm/Group | Part B: Moxifloxacin 400 mg
Number analyzed (Participants) | 60
ms
  0.25 hours post-dose | 2.2 [0.89 to 3.53]
  0.5 hours post-dose | 8.6 [7.11 to 10.05]
  0.75 hours post-dose | 10.1 [8.51 to 11.67]
  1 hour post-dose | 10.2 [8.74 to 11.58]
  1.5 hours post-dose | 11.1 [9.61 to 12.59]
  2 hours post-dose | 12.7 [11.13 to 14.17]
  3 hours post-dose | 13.1 [11.71 to 14.57]
  4 hours post-dose | 12.9 [11.37 to 14.42]
  8 hours post-dose | 9.7 [7.75 to 11.62]
  12 hours post-dose | 9.0 [6.85 to 11.06]
  24 hours post-dose | 5.3 [3.78 to 6.76]

10. Secondary Outcome: Change From Baseline in Heart Rate After Omecamtiv Mecarbil Dosing in Part B
Description: Change from baseline in heart rate (HR) was calculated based on a linear mixed-effects model with period, sequence, time (categorical), treatment, and time-by-treatment interaction as fixed effects and baseline HR as a covariate.
Time Frame: Baseline (average of samples taken at -1.25, -1, and -0.75 hours predose on day 1 of the OM treatment period) and at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 8, 12, and 24 hours post-dose.
Population: The QT/QTc analysis set
Measure: Least Squares Mean (90% Confidence Interval); unit: bpm
Arm/Group | Part B: Omecamtiv Mecarbil 50 mg
Number analyzed (Participants) | 60
bpm
  0.25 hours post-dose | 1.3 [0.37 to 2.16]
  0.5 hours post-dose | 1.2 [0.38 to 2.12]
  0.75 hours post-dose | 1.4 [0.51 to 2.37]
  1 hour post-dose | 0.2 [-0.86 to 1.18]
  1.5 hours post-dose | -0.5 [-1.44 to 0.46]
  2 hours post-dose | -0.2 [-1.10 to 0.77]
  3 hours post-dose | 1.1 [0.09 to 2.09]
  4 hours post-dose | 1.8 [0.77 to 2.84]
  8 hours post-dose | 7.8 [6.57 to 9.11]
  12 hours post-dose | 8.3 [7.07 to 9.55]
  24 hours post-dose | 2.8 [1.66 to 3.95]

11. Secondary Outcome: Change From Baseline in QTcF After Omecamtiv Mecarbil Dosing in Part B
Description: Change from baseline in QTcF was calculated based on a linear mixed-effects model with period, sequence, time (categorical), treatment, and time-by-treatment interaction as fixed effects and baseline QTcF as a covariate.
Time Frame: as for outcome 10
Population: The QT/QTc analysis set
Measure: Least Squares Mean (90% Confidence Interval); unit: ms
Arm/Group | Part B: Omecamtiv Mecarbil 50 mg
Number analyzed (Participants) | 60
ms
  0.25 hours post-dose | -6.3 [-7.38 to -5.25]
  0.5 hours post-dose | -9.1 [-10.30 to -7.98]
  0.75 hours post-dose | -8.6 [-9.84 to -7.38]
  1 hour post-dose | -8.1 [-9.23 to -6.99]
  1.5 hours post-dose | -5.5 [-6.66 to -4.33]
  2 hours post-dose | -5.2 [-6.40 to -4.02]
  3 hours post-dose | -4.9 [-6.04 to -3.78]
  4 hours post-dose | -3.3 [-4.51 to -2.12]
  8 hours post-dose | -7.1 [-8.55 to -5.64]
  12 hours post-dose | -6.6 [-8.18 to -5.04]
  24 hours post-dose | -4.1 [-5.23 to -2.89]

12. Secondary Outcome: Change From Baseline in PR Interval After Omecamtiv Mecarbil Dosing in Part B
Description: The PR interval is the time from the onset of the P-wave to the start of the next QRS complex. Change from baseline was calculated based on a linear mixed-effects model with period, sequence, time (categorical), treatment, and time-by-treatment interaction as fixed effects and baseline PR interval as covariate.
Time Frame: as for outcome 10
Population: The QT/QTc analysis set
Measure: Least Squares Mean (90% Confidence Interval); unit: ms
Arm/Group | Part B: Omecamtiv Mecarbil 50 mg
Number analyzed (Participants) | 60
ms
  0.25 hours post-dose | -0.5 [-1.76 to 0.67]
  0.5 hours post-dose | 1.0 [-0.20 to 2.24]
  0.75 hours post-dose | 0.4 [-0.87 to 1.76]
  1 hour post-dose | 0.4 [-1.02 to 1.75]
  1.5 hours post-dose | -1.2 [-2.40 to -0.08]
  2 hours post-dose | -0.8 [-2.16 to 0.60]
  3 hours post-dose | -2.0 [-3.37 to -0.67]
  4 hours post-dose | -3.2 [-4.64 to -1.77]
  8 hours post-dose | -7.5 [-9.28 to -5.67]
  12 hours post-dose | -7.8 [-9.69 to -5.96]
  24 hours post-dose | -2.1 [-3.71 to -0.58]

13. Secondary Outcome: Change From Baseline in QRS After Omecamtiv Mecarbil Dosing in Part B
Description: The QRS complex is a combination of the Q wave, R wave and S wave on an ECG tracing, and represents ventricular depolarization. Change from baseline was calculated based on a linear mixed-effects model with period, sequence, time (categorical), treatment, and time-by-treatment interaction as fixed effects and baseline QRS as covariate.
Time Frame: as for outcome 10
Population: The QT/QTc analysis set
Measure: Least Squares Mean (90% Confidence Interval); unit: ms
Arm/Group | Part B: Omecamtiv Mecarbil 50 mg
Number analyzed (Participants) | 60
ms
  0.25 hours post-dose | -0.2 [-0.42 to -0.01]
  0.5 hours post-dose | 0.0 [-0.28 to 0.22]
  0.75 hours post-dose | -0.2 [-0.37 to 0.02]
  1 hour post-dose | 0.0 [-0.28 to 0.33]
  1.5 hours post-dose | -0.2 [-0.41 to 0.06]
  2 hours post-dose | -0.3 [-0.51 to -0.02]
  3 hours post-dose | 0.00 [-0.26 to 0.18]
  4 hours post-dose | 0.1 [-0.14 to 0.34]
  8 hours post-dose | -0.4 [-0.80 to 0.03]
  12 hours post-dose | -0.7 [-1.03 to -0.32]
  24 hours post-dose | -0.3 [-0.61 to 0.08]

14. Secondary Outcome: Slope of Omecamtiv Mecarbil Plasma Concentration Estimated From Concentration-QTc Analysis in Part B
Description: The relationship between omecamtiv mecarbil plasma concentration and ΔQTcF was investigated by linear mixed-effects modeling with ΔQTcF as the dependent variable, time-matched concentration of OM as the explanatory variable (0 for placebo), centered baseline QTcF (i.e., baseline QTcF for individual subject minus the population mean baseline QTcF for all subjects in the same period) as an additional covariate, study treatment (OM = 1 or placebo = 0) and time (i.e., post-dose time point) as fixed effects, and a random intercept and slope per subject. From the model, the slope (i.e., the regression parameter for the concentration) was estimated together with the 2-sided 90% CI.
Time Frame: as for outcome 10
Population: The PK/QTc analysis set included all participants who were in both the QT/QTc and PK analysis sets with at least 1 pair of post-dose PK and QTcF data from the same timepoint.
Measure: Number (90% Confidence Interval); unit: ms per ng/mL
Arm/Group | Part B: Omecamtiv Mecarbil 50 mg
Number analyzed (Participants) | 60
ms per ng/mL | -0.011 [-0.0154 to -0.0073]

15. Secondary Outcome: Placebo-corrected Change From Baseline in Heart Rate After Omecamtiv Mecarbil Dosing in Part B
Description: Change from baseline in heart rate (ΔHR) was calculated based on a linear mixed-effects model with period, sequence, time (categorical), treatment, and time-by-treatment interaction as fixed effects and baseline HR as covariate.
  Placebo-corrected ΔHR (ΔΔHR) was calculated as the adjusted mean ΔHR after OM dosing minus adjusted mean ΔHR after placebo dosing.
Time Frame: as for outcome 10
Population: The QT/QTc analysis set
Measure: Least Squares Mean (90% Confidence Interval); unit: bpm
Arm/Group | Part B: Omecamtiv Mecarbil 50 mg
Number analyzed (Participants) | 60
bpm
  0.25 hours post-dose | -0.9 [-1.84 to 0.09]
  0.5 hours post-dose | -1.3 [-2.27 to -0.42]
  0.75 hours post-dose | -0.6 [-1.68 to 0.40]
  1 hour post-dose | -2.3 [-3.54 to -1.15]
  1.5 hours post-dose | -1.9 [-2.93 to -0.78]
  2 hours post-dose | -1.5 [-2.57 to -0.47]
  3 hours post-dose | -0.9 [-2.02 to 0.30]
  4 hours post-dose | 0.5 [-0.71 to 1.74]
  8 hours post-dose | -0.1 [-1.72 to 1.49]
  12 hours post-dose | -1.0 [-2.57 to 0.55]
  24 hours post-dose | -1.7 [-3.09 to -0.28]

16. Secondary Outcome: Placebo-corrected Change From Baseline in PR Interval After Omecamtiv Mecarbil Dosing in Part B
Description: Change from baseline in PR interval (ΔPR) was calculated based on a linear mixed-effects model with period, sequence, time (categorical), treatment, and time-by-treatment interaction as fixed effects and baseline PR interval as covariate.
  Placebo-corrected ΔPR (ΔΔPR) was calculated as the adjusted mean ΔPR after OM dosing minus adjusted mean ΔPR after placebo dosing.
Time Frame: as for outcome 10
Population: The QT/QTc analysis set
Measure: Least Squares Mean (90% Confidence Interval); unit: ms
Arm/Group | Part B: Omecamtiv Mecarbil 50 mg
Number analyzed (Participants) | 60
ms
  0.25 hours post-dose | 0.6 [-1.02 to 2.26]
  0.5 hours post-dose | 0.9 [-0.74 to 2.54]
  0.75 hours post-dose | -0.3 [-2.07 to 1.50]
  1 hour post-dose | 1.0 [-0.89 to 2.87]
  1.5 hours post-dose | 0.1 [-1.46 to 1.64]
  2 hours post-dose | 1.9 [-0.02 to 3.74]
  3 hours post-dose | 0.4 [-1.41 to 2.26]
  4 hours post-dose | 0.1 [-1.83 to 2.09]
  8 hours post-dose | -1.6 [-4.12 to 0.88]
  12 hours post-dose | -1.0 [-3.57 to 1.61]
  24 hours post-dose | -0.1 [-2.22 to 2.08]

17. Secondary Outcome: Placebo-corrected Change From Baseline in QRS After Omecamtiv Mecarbil Dosing in Part B
Description: Change from baseline in QRS (ΔQRS) was calculated based on a linear mixed-effects model with period, sequence, time (categorical), treatment, and time-by-treatment interaction as fixed effects and baseline QRS as covariate.
  Placebo-corrected ΔQRS (ΔΔQRS) was calculated as the adjusted mean ΔQRS after OM dosing minus adjusted mean ΔQRS after placebo dosing.
Time Frame: as for outcome 10
Population: The QT/QTc analysis set
Measure: Least Squares Mean (90% Confidence Interval); unit: ms
Arm/Group | Part B: Omecamtiv Mecarbil 50 mg
Number analyzed (Participants) | 60
ms
  0.25 hours post-dose | -0.1 [-0.34 to 0.21]
  0.5 hours post-dose | -0.1 [-0.41 to 0.28]
  0.75 hours post-dose | -0.1 [-0.33 to 0.20]
  1 hour post-dose | -0.1 [-0.53 to 0.32]
  1.5 hours post-dose | 0.0 [-0.33 to 0.32]
  2 hours post-dose | 0.1 [-0.28 to 0.39]
  3 hours post-dose | 0.1 [-0.18 to 0.41]
  4 hours post-dose | 0.1 [-0.22 to 0.44]
  8 hours post-dose | 0.3 [-0.32 to 0.85]
  12 hours post-dose | 0.4 [-0.07 to 0.91]
  24 hours post-dose | -0.1 [-0.60 to 0.36]

18. Secondary Outcome: Number of Participants With Recorded Outlier Values for QTcF, HR, PR, and QRS After Omecamtiv Mecarbil Dosing in Part B
Description: Outliers were predefined according to the following categories:
  QTcF:
  Treatment-emergent value of > 450 and ≤ 480 ms when not present at baseline (new onset) Treatment-emergent value of > 480 and ≤ 500 ms when not present at baseline (new onset) Treatment-emergent value of > 500 ms when not present at baseline (new onset) Increase of QTcF from baseline of > 30 and ≤ 60 ms Increase of QTcF from baseline > 60 ms Increase of PR from baseline > 25% resulting in PR > 200 ms Increase of QRS from baseline > 25% resulting in QRS > 120 ms Decrease of HR from baseline > 25% resulting in HR < 50 bpm Increase of HR from baseline > 25% resulting in HR > 100 bpm
Time Frame: Day 1 of the OM treatment period at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 8, 12, and 24 hours post-dose.
Population: QT/QTc analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Omecamtiv Mecarbil 50 mg
Number analyzed (Participants) | 60
Participants
  QTcF > 450 and ≤ 480 ms (new onset) | 1
  QTcF > 480 and ≤ 500 ms (new onset) | 0
  QTcF > 500 ms (new onset) | 0
  Increase in ΔQTcF > 30 and ≤ 60 ms | 0
  Increase in ΔQTcF > 60 ms | 0
  HR < 50 bpm with a decrease in ΔHR > 25% | 0
  HR > 100 bpm with an increase in ΔHR > 25% | 0
  PR > 200 ms with an increase in ΔPR > 25% | 0
  QRS > 120 ms with an increase in ΔQRS > 25% | 0

19. Secondary Outcome: Number of Participants With Treatment-emergent Changes in T-wave Morphology and U-wave Presence After Omecamtiv Mecarbil Dosing in Part B
Description: T-wave abnormalities were categorized as follows:
  Flat T-wave: T amplitude < 1 mm (either positive or negative) including flat isoelectric line Notched T-wave (+): Presence of notch(es) of at least 0.05 mV amplitude on ascending or descending arm of the positive T-wave Biphasic: T-wave that contains a second component with an opposite phase that is at least 0.1 mV deep (both positive/negative and negative/positive and polyphasic T-waves included) Normal T-wave (-): T amplitude that is negative, without biphasic T-wave or notches Notched T-wave (-): Presence of notch(es) of at least 0.05 mV amplitude on descending or ascending arm of the negative T-wave U waves: Presence of abnormal U-waves
Time Frame: Day 1 of the OM treatment period at 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 8, 12, and 24 hours post-dose.
Population: QT/QTc analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Omecamtiv Mecarbil 50 mg
Number analyzed (Participants) | 60
Participants
  Flat T-wave | 0
  Notched T-wave (+) | 0
  Biphasic T-wave | 0
  Normal T-wave (-) | 0
  Notched T-wave (-) | 0
  U-Wave presence | 0

20. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: A TEAE was defined as an adverse event (AE) that started during or after the first dose, or started prior to the first dose and increased in severity after the first dose. A treatment-related TEAE was defined as a TEAE with a relationship of related to the study treatment as determined by the investigator.
  The Investigator assessed the severity of each AE reported during the study based on the following grading scale:
  Mild: Aware of sign or symptom, easily tolerated Moderate: Discomfort enough to cause interference with usual activity Severe: Incapacitating, inability to work or do usual activity
  SAEs were defined as any untoward medical occurrence that met at least 1 of the following serious criteria:
  * Resulted in Death
  * Was life-threatening
  * Required in-patient hospitalization or prolongation of existing hospitalization
  * Resulted in persistent or significant disability/incapacity
  * Was a congenital anomaly/birth defect
  * Other medically important serious event
Time Frame: From first dose of study treatment to day 6 of each treatment period
Population: The safety population included all participants who received at least 1 dose of study treatment (OM, placebo, or moxifloxacin) and had at least 1 postdose safety assessment.
Measure: Count of Participants; unit: Participants
Groups:
- Part A: Omecamtiv Mecarbil 25 mg: After an overnight fast of at least 10 hours participants received a single oral dose of 25 mg omecamtiv mecarbil on Day 1.
- Part B: Placebo: Participants received a single oral dose of placebo on day 1 of treatment period 1, 2, or 3, depending on sequence assignment.
Arm/Group | Part A: Omecamtiv Mecarbil 25 mg | Part B: Placebo | Part B: Omecamtiv Mecarbil 50 mg | Part B: Moxifloxacin 400 mg
Number analyzed (Participants) | 70 | 60 | 60 | 60
Participants
  Any TEAE | 20 | 26 | 24 | 29
  Serious TEAE | 0 | 0 | 0 | 0
  TEAE leading to discontinuation | 0 | 0 | 0 | 0
  TEAE leading to death | 0 | 0 | 0 | 0
  Mild TEAE | 19 | 25 | 24 | 28
  Moderate TEAE | 2 | 1 | 1 | 2
  Severe TEAE | 0 | 0 | 0 | 0
  Treatment-related TEAE | 2 | 0 | 4 | 2
  Treatment-related serious TEAE | 0 | 0 | 0 | 0
  Treatment-related TEAE leading to discontinuation | 0 | 0 | 0 | 0
  Treatment-related TEAE leading to death | 0 | 0 | 0 | 0
  Treatment-related mild TEAE | 2 | 0 | 4 | 2
  Treatment-related moderate TEAE | 0 | 0 | 0 | 0
  Treatment-related severe TEAE | 0 | 0 | 0 | 0

21. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Vital Signs, Laboratory Tests, or Electrocardiogram Findings
Description: Blood and urine samples were collected for clinical laboratory evaluations (including clinical chemistry, hematology, urinalysis, and serology). Vital signs included blood pressure, pulse rate and body temperature. Standard safety 12-lead ECGs were recorded after the subject had been supine or semi-recumbent and at rest for at least 5 minutes to detect any immediate ECG effects for subject safety. These ECGs were viewed locally. The Investigator determined whether an abnormal value in an individual participant represented a clinically significant change from the participant's baseline values.
Time Frame: From first dose up to day 6 of each treatment period
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Omecamtiv Mecarbil 25 mg | Part B: Placebo | Part B: Omecamtiv Mecarbil 50 mg | Part B: Moxifloxacin 400 mg
Number analyzed (Participants) | 70 | 60 | 60 | 60
Participants
  Clinical Laboratory Evaluations | 0 | 0 | 0 | 0
  Vital Signs | 0 | 0 | 0 | 0
  12-lead Electrocardiogram | 0 | 0 | 0 | 0

22. Post Hoc Outcome: Change From Baseline in QTcF After Each Treatment In Part 2
Description: as for outcome 11
Time Frame: as for outcome 10
Population: The QT/QTc analysis set
Measure: Least Squares Mean (90% Confidence Interval); unit: ms
Arm/Group | Part B: Omecamtiv Mecarbil 50 mg | Part B: Moxifloxacin 400 mg | Part B: Placebo
Number analyzed (Participants) | 60 | 60 | 60
ms
  0.25 hours post-dose | -6.3 [-7.38 to -5.25] | -1.6 [-2.61 to -0.49] | -3.8 [-4.82 to -2.70]
  0.5 hours post-dose | -9.1 [-10.30 to -7.98] | 4.4 [3.21 to 5.53] | -4.2 [-5.37 to -3.05]
  0.75 hours post-dose | -8.6 [-9.84 to -7.38] | 7.2 [6.01 to 8.47] | -2.8 [-4.08 to -1.62]
  1 hour post-dose | -8.1 [-9.23 to -6.99] | 8.8 [7.63 to 9.88] | -1.4 [-2.52 to -0.28]
  1.5 hours post-dose: number analyzed (Participants) | 60 | 59 | 60
  1.5 hours post-dose | -5.5 [-6.66 to -4.33] | 10.1 [8.89 to 11.23] | -1.0 [-2.20 to 0.13]
  2 hours post-dose | -5.2 [-6.40 to -4.02] | 10.1 [8.95 to 11.33] | -2.5 [-3.70 to -1.33]
  3 hours post-dose | -4.9 [-6.04 to -3.78] | 9.8 [8.63 to 10.89] | -3.4 [-4.51 to -2.25]
  4 hours post-dose | -3.3 [-4.51 to -2.12] | 10.4 [9.21 to 11.59] | -2.5 [-3.68 to -1.30]
  8 hours post-dose: number analyzed (Participants) | 60 | 59 | 60
  8 hours post-dose | -7.1 [-8.55 to -5.64] | 4.8 [3.30 to 6.22] | -4.9 [-6.38 to -3.47]
  12 hours post-dose | -6.6 [-8.18 to -5.04] | 4.2 [2.66 to 5.80] | -4.7 [-6.30 to -3.16]
  24 hours post-dose | -4.1 [-5.23 to -2.89] | 2.4 [1.23 to 3.57] | -2.9 [-4.04 to -1.70]

23. Post Hoc Outcome: Change From Baseline in Heart Rate After Each Treatment In Part 2
Description: as for outcome 10
Time Frame: as for outcome 10
Population: The QT/QTc analysis set
Measure: Least Squares Mean (90% Confidence Interval); unit: bpm
Arm/Group | Part B: Omecamtiv Mecarbil 50 mg | Part B: Moxifloxacin 400 mg | Part B: Placebo
Number analyzed (Participants) | 60 | 60 | 60
bpm
  0.25 hours post-dose | 1.3 [0.37 to 2.16] | 2.1 [1.22 to 3.01] | 2.1 [1.25 to 3.04]
  0.5 hours post-dose | 1.2 [0.38 to 2.12] | 4.0 [3.14 to 4.88] | 2.6 [1.72 to 3.47]
  0.75 hours post-dose | 1.4 [0.51 to 2.37] | 5.3 [4.33 to 6.20] | 2.1 [1.15 to 3.01]
  1 hour post-dose | 0.2 [-0.86 to 1.18] | 5.4 [4.39 to 6.43] | 2.5 [1.49 to 3.53]
  1.5 hours post-dose: number analyzed (Participants) | 60 | 59 | 60
  1.5 hours post-dose | -0.5 [-1.44 to 0.46] | 2.0 [1.06 to 2.97] | 1.4 [0.41 to 2.32]
  2 hours post-dose | -0.2 [-1.10 to 0.77] | 2.0 [1.05 to 2.93] | 1.4 [0.41 to 2.29]
  3 hours post-dose | 1.1 [0.09 to 2.09] | 3.0 [1.97 to 3.97] | 2.0 [0.96 to 2.95]
  4 hours post-dose | 1.8 [0.77 to 2.84] | 2.9 [1.88 to 3.95] | 1.3 [0.25 to 2.32]
  8 hours post-dose: number analyzed (Participants) | 60 | 59 | 60
  8 hours post-dose | 7.8 [6.57 to 9.11] | 9.1 [7.83 to 10.38] | 8.0 [6.69 to 9.22]
  12 hours post-dose | 8.3 [7.07 to 9.55] | 9.6 [8.37 to 10.85] | 9.3 [8.08 to 10.56]
  24 hours post-dose | 2.8 [1.66 to 3.95] | 3.4 [2.30 to 4.59] | 4.5 [3.34 to 5.63]

24. Post Hoc Outcome: Change From Baseline in PR Interval After Each Treatment In Part 2
Description: as for outcome 12
Time Frame: as for outcome 10
Population: The QT/QTc analysis set
Measure: Least Squares Mean (90% Confidence Interval); unit: ms
Arm/Group | Part B: Omecamtiv Mecarbil 50 mg | Part B: Moxifloxacin 400 mg | Part B: Placebo
Number analyzed (Participants) | 60 | 60 | 60
ms
  0.25 hours post-dose | -0.5 [-1.76 to 0.67] | -1.6 [-2.85 to -0.42] | -1.2 [-2.38 to 0.06]
  0.5 hours post-dose | 1.0 [-0.20 to 2.24] | -0.6 [-1.78 to 0.66] | 0.1 [-1.10 to 1.34]
  0.75 hours post-dose | 0.4 [-0.87 to 1.76] | -1.1 [-2.40 to 0.24] | 0.7 [-0.58 to 2.05]
  1 hour post-dose | 0.4 [-1.02 to 1.75] | -1.5 [-2.83 to -0.07] | -0.6 [-2.00 to 0.76]
  1.5 hours post-dose: number analyzed (Participants) | 60 | 59 | 60
  1.5 hours post-dose | -1.2 [-2.40 to -0.08] | -2.1 [-3.24 to -0.91] | -1.3 [-2.48 to -0.17]
  2 hours post-dose | -0.8 [-2.16 to 0.60] | -1.6 [-2.99 to -0.24] | -2.6 [-4.02 to -1.26]
  3 hours post-dose | -2.0 [-3.37 to -0.67] | -3.3 [-4.64 to -1.94] | -2.5 [-3.80 to -1.10]
  4 hours post-dose | -3.2 [-4.64 to -1.77] | -4.5 [-5.90 to -3.04] | -3.3 [-4.77 to -1.90]
  8 hours post-dose: number analyzed (Participants) | 60 | 59 | 60
  8 hours post-dose | -7.5 [-9.28 to -5.67] | -7.7 [-9.55 to -5.93] | -5.8 [-7.65 to -4.04]
  12 hours post-dose | -7.8 [-9.69 to -5.96] | -7.5 [-9.37 to -5.63] | -6.8 [-8.72 to -4.98]
  24 hours post-dose | -2.1 [-3.71 to -0.58] | -2.6 [-4.14 to -1.01] | -2.1 [-3.64 to -0.51]

25. Post Hoc Outcome: Change From Baseline in QRS After Each Treatment In Part 2
Description: as for outcome 13
Time Frame: as for outcome 10
Population: The QT/QTc analysis set
Measure: Least Squares Mean (90% Confidence Interval); unit: ms
Arm/Group | Part B: Omecamtiv Mecarbil 50 mg | Part B: Moxifloxacin 400 mg | Part B: Placebo
Number analyzed (Participants) | 60 | 60 | 60
ms
  0.25 hours post-dose | -0.2 [-0.42 to -0.01] | -0.2 [-0.43 to -0.02] | -0.2 [-0.36 to 0.05]
  0.5 hours post-dose | 0.0 [-0.28 to 0.22] | -0.1 [-0.36 to 0.15] | 0.0 [-0.22 to 0.29]
  0.75 hours post-dose | -0.2 [-0.37 to 0.02] | 0.0 [-0.18 to 0.21] | -0.1 [-0.31 to 0.08]
  1 hour post-dose | 0.0 [-0.28 to 0.33] | 0.1 [-0.25 to 0.36] | 0.1 [-0.18 to 0.44]
  1.5 hours post-dose: number analyzed (Participants) | 60 | 59 | 60
  1.5 hours post-dose | -0.2 [-0.41 to 0.06] | 0.0 [-0.27 to 0.21] | -0.2 [-0.41 to 0.07]
  2 hours post-dose | -0.3 [-0.51 to -0.02] | 0.1 [-0.16 to 0.33] | -0.3 [-0.56 to -0.07]
  3 hours post-dose | 0.00 [-0.26 to 0.18] | 0.1 [-0.15 to 0.29] | -0.2 [-0.37 to 0.07]
  4 hours post-dose | 0.1 [-0.14 to 0.34] | 0.2 [-0.04 to 0.44] | 0.0 [-0.25 to 0.23]
  8 hours post-dose: number analyzed (Participants) | 60 | 59 | 60
  8 hours post-dose | -0.4 [-0.80 to 0.03] | -0.3 [-0.76 to 0.08] | -0.6 [-1.07 to -0.23]
  12 hours post-dose | -0.7 [-1.03 to -0.32] | -0.7 [-1.10 to -0.40] | -1.1 [-1.45 to -0.74]
  24 hours post-dose | -0.3 [-0.61 to 0.08] | 0.0 [-0.35 to 0.33] | -0.1 [-0.49 to 0.20]

ADVERSE EVENTS:
Time Frame: From first dose of study drug to 6 days post-dose in each treatment period.
Groups:
- Overall: ALL TREATED SUBJECTS
Arm/Group | Part A: Omecamtiv Mecarbil 25 mg | Part B: Placebo | Part B: Omecamtiv Mecarbil 50 mg | Part B: Moxifloxacin 400 mg | Overall
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/60 | 0/60 | 0/60 | 0/70
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/60 | 0/60 | 0/60 | 0/70
Other Adverse Events (participants affected / at risk) | 14/70 | 16/60 | 13/60 | 18/60 | 39/70
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Omecamtiv Mecarbil 25 mg (N=70) | Part B: Placebo (N=60) | Part B: Omecamtiv Mecarbil 50 mg (N=60) | Part B: Moxifloxacin 400 mg (N=60) | Overall (N=70)
Nausea (Gastrointestinal disorders) | 1 | 4 | 1 | 3 | 7
Nasopharyngitis (Infections and infestations) | 1 | 1 | 2 | 0 | 4
Post procedural complication (Injury, poisoning and procedural complications) | 4 | 2 | 3 | 1 | 10
Post procedural erythema (Injury, poisoning and procedural complications) | 2 | 6 | 5 | 5 | 15
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 3 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3 | 3
Dizziness (Nervous system disorders) | 1 | 2 | 0 | 2 | 5
Headache (Nervous system disorders) | 1 | 3 | 3 | 2 | 9
Insomnia (Psychiatric disorders) | 1 | 2 | 2 | 1 | 6
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 2 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 3 | 1 | 7
Rash (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 1 | 4
Rash papular (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2019-08-23): https://cdn.clinicaltrials.gov/large-docs/08/NCT04175808/Prot_000.pdf
  • Statistical Analysis Plan: SAP Version 1 (2019-12-10): https://cdn.clinicaltrials.gov/large-docs/08/NCT04175808/SAP_001.pdf